CLINICAL TRIAL: NCT04837768
Title: Effect of Intramuscular Progesterone Supplementation on Clinical and Ongoing Pregnancy Rates in Patients With Low Serum Progesterone Levels on the Day of Embryo Transfer in Artificial Frozen Cycles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdelfatah Mohamed Kamel Eldesouky, Assistant Lecturer in the Department of Obstetrics and Gynecology, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Progesterone in HRT FET cycles
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Serum Progesterone Levels; Progesterone Supplementation; Frozen Embryo Transfer; Clinical Pregnancy Rates; Ongoing Pregnancy Rates

STUDY DESIGN:
Intervention Model Description: Patients undergoing frozen cycles following ICSI will receive artificial endometrial preparation from day 2/3 of their cycle in the form of 2mg Estradiol Valerate pills thrice daily for 7-10 days. After confirming endometrial thickness > 7mm via TVS, progesterone supplementation will start via Prontogest® 400mg vaginal pessaries twice daily for 5 days, ending with the day of embryo transfer (ET).
  On the morning of ET, serum progesterone will be measured and if the value is over 9.2ng/ml, only the traditional twice daily vaginal progesterone will be resumed until 12 weeks gestation. If the value is under 9.2 ng/ml, intramuscular progesterone supplementation with Prontogest® 100mg will be added in twice-weekly doses (every 3 days) to the vaginal supplementation.
  Quantitative β-hcg 2 weeks after ET to detect chemical pregnancies. Ultrasound 4 weeks after ET to detect clinical pregnancies. Ultrasound repeated at 12 weeks to confirm ongoing pregnancy rates.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serum Progesterone Levels >9.2 ng/ml (Active Comparator): These patients will receive only twice-daily vaginal progesterone supplementation following embryo transfer
  Interventions: Drug: Twice-daily transvaginal progesterone supplementation
- Serum Progesterone Levels <9.2 ng/ml (Active Comparator): These patients will receive twice-weekly intramuscular progesterone supplementation in addition to the twice-daily vaginal supplementation following embryo transfer
  Interventions: Drug: Twice-weekly intramuscular + Twice-daily transvaginal progesterone supplementation

INTERVENTIONS:
Drug: Twice-daily transvaginal progesterone supplementation — Patients with serum progesterone levels >9.2 ng/ml on the day of embryo transfer in artificial frozen cycles will receive the traditional twice-daily vaginal progesterone supplementation till 12 weeks gestation.
  Arms: Serum Progesterone Levels >9.2 ng/ml
Drug: Twice-weekly intramuscular + Twice-daily transvaginal progesterone supplementation — Patients with serum progesterone levels <9.2 ng/ml on the day of embryo transfer in artificial frozen cycles will receive the twice-daily vaginal progesterone in addition to twice-weekly intramuscular progesterone supplementation till 12 weeks gestation.
  Arms: Serum Progesterone Levels <9.2 ng/ml

SUMMARY:
The aim of this study is to investigate whether intramuscular progesterone supplementation will improve clinical pregnancy rates and ongoing pregnancy rates in patients with decreased serum progesterone levels on the day of embryo transfer in artificial frozen cycles.

DETAILED DESCRIPTION:
Cryopreservation of frozen-thawed embryos has become a cardinal procedure in assisted reproductive therapies. This can be attributed to the development of the vitrification process and the improvement of embryo survival rates after thawing, leading to the progressive increase in the use of frozen embryo transfer (FET).

The need for FET has also increased greatly due to the implementation of a single embryo transfer policy in many areas of the world to reduce multiple pregnancies. This has led to an increase in surplus embryos derived from ovarian stimulation cycles. Moreover, although the 'freeze all' technique or elective embryo cryopreservation was mainly developed for patients with an increased risk of developing ovarian hyperstimulation syndrome, its use has now been extended to cover other indications, such as cycles involving pre-implantation genetic diagnosis, late-follicular progesterone elevation and embryo-endometrial asynchrony.

Despite this increased need for FET, there still exists debate over the best method to implement the practice. The two most common used treatment regimens to prepare the endometrium for embryo transfer are the so-called natural cycle (NC) and the hormone replacement therapy (HRT) cycle.

In a NC FET, there is no medical intervention apart from ultrasound monitoring during the proliferative phase, to schedule the transfer when the endometrium is synchronized to the developmental stage of the embryo. Although the advantage is the absence of estrogen supplementation, this protocol entails more frequent visits to the clinic and less cycle control. Despite this, there is still an ongoing debate whether frozen embryos transferred in a 'more physiologic' non-stimulated endometrium, may not only result in higher pregnancy rates, but also potentially decrease maternal and neonatal morbidity.

On the other hand, in the HRT cycle, also referred to as an artificial cycle, exogenous administration of estrogens and progesterone is used to mimic a natural cycle and therefore endometrial development. Although originally developed to allow embryo transfers in recipients of donated oocytes, the HRT protocol has proven to be successful in the general population as well.

The advantage of this protocol is the easy scheduling and minimal cycle monitoring. There are however, potential disadvantages associated with its widespread usage, including the increased expense and risks of estrogen supplementation such as thromboembolic events.

Generally speaking, in HRT cycles, progesterone supplementation begins once the proliferation of the endometrium with the administration of estrogens is considered sufficient. Progesterone is initiated to promote the final phase of endometrial preparation prior to embryo transfer, however, there is little agreement on the ideal route or dose of progesterone supplementation itself.

As regards the route of administration, when compared to intramuscular (IM) injections, patients seem to prefer the vaginal route owing to its quick, easy and painless administration. Despite this, there is limited data comparing IM versus vaginal progesterone administration, with some being in favour of the IM route and others showing no significant differences in terms of outcome.

However, the more recent focus on intramuscular rather than the traditional transvaginal progesterone supplementation, stems from newer mounting evidence that transvaginal supplementation not only increases vaginal discharge, but also has a limited effect in increasing serum progesterone levels.

Boynukalin et al., 2019 explored the idea of intramuscular progesterone supplementation in HRT FET cycles further, by substituting the traditional vaginal progesterone with 100mg of daily IM progesterone during endometrial preparation and thereafter till the 10th week of pregnancy. They found that the mean progesterone level on the day of ET was significantly higher in patients who later had an ongoing pregnancy (28 ng/ml) than those who did not have an ongoing pregnancy (16.4 ng/ml) with a p-value of 0.039. They did however conclude, that further investigation is needed for the individualization of intramuscular progesterone doses to reach optimal pregnancy rates.

Thus, more attention has been given recently to measuring serum progesterone during HRT FET cycles. Kofinas et al., 2015 suggested that progesterone levels >20 ng/ml (possibly due to an escape ovulation and subsequent embryo-endometrial asynchrony) on the day of transfer have been associated with decreased ongoing pregnancy and live birth rates. On the other hand, Yovich, et al., 2015 proposed an optimal mid-luteal progesterone range between 22 and 31 ng/ml.

Most recently, Labarta et al., 2017 investigated the relationship between serum progesterone levels on the day of embryo transfer (ET) and ongoing pregnancy rate (OPR). Their study recommended a minimum serum progesterone threshold (9.2 ng/ml) to optimize OPR in artificial cycles using transvaginal progesterone and this value could theoretically be used to decide if ET should be postponed or not.

Extrapolating from this data, we intend to investigate whether intramuscular progesterone supplementation can help improve OPR rates in the aforementioned patients with decreased serum progesterone on the day of ET. In other words, we intend to investigate further the concept of individualizing luteal phase support in HRT FET cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Age range 20-40 years
2. BMI < 40 kg/m2
3. Endometrial thickness >7mm
4. Double embryo transfer (Day 5), Grade 1 or 2.

Exclusion Criteria:

1. Autoimmune diseases
2. Uncontrolled medical conditions
3. Recurrent implantation failure
4. Anatomical uterine abnormalities as polyps, fibroids or Müllerian anomalies.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 354 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rates | 4 weeks after the day of embryo transfer
  Detected via ultrasound

SECONDARY OUTCOMES:
Ongoing pregnancy rates | 12 weeks after the day of embryo transfer
  Detected via ultrasound

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Cairo University, Faculty of Medicine, Department of Obstetrics and Gynecology, Cairo
  - AlBoshra IVF & Infertility Treatment Centre, Cairo

REFERENCES:
- [Background] Labarta E, Mariani G, Holtmann N, Celada P, Remohi J, Bosch E. Low serum progesterone on the day of embryo transfer is associated with a diminished ongoing pregnancy rate in oocyte donation cycles after artificial endometrial preparation: a prospective study. Hum Reprod. 2017 Dec 1;32(12):2437-2442. doi: 10.1093/humrep/dex316. PMID 29040638
- [Background] Boynukalin FK, Gultomruk M, Turgut E, Demir B, Findikli N, Serdarogullari M, Coban O, Yarkiner Z, Bahceci M. Measuring the serum progesterone level on the day of transfer can be an additional tool to maximize ongoing pregnancies in single euploid frozen blastocyst transfers. Reprod Biol Endocrinol. 2019 Nov 29;17(1):102. doi: 10.1186/s12958-019-0549-9. PMID 31783865
- [Background] Kofinas JD, Blakemore J, McCulloh DH, Grifo J. Serum progesterone levels greater than 20 ng/dl on day of embryo transfer are associated with lower live birth and higher pregnancy loss rates. J Assist Reprod Genet. 2015 Sep;32(9):1395-9. doi: 10.1007/s10815-015-0546-7. Epub 2015 Aug 4. PMID 26238390
- [Background] Yovich JL, Conceicao JL, Stanger JD, Hinchliffe PM, Keane KN. Mid-luteal serum progesterone concentrations govern implantation rates for cryopreserved embryo transfers conducted under hormone replacement. Reprod Biomed Online. 2015 Aug;31(2):180-91. doi: 10.1016/j.rbmo.2015.05.005. Epub 2015 May 18. PMID 26099447
- [Background] Mackens S, Santos-Ribeiro S, van de Vijver A, Racca A, Van Landuyt L, Tournaye H, Blockeel C. Frozen embryo transfer: a review on the optimal endometrial preparation and timing. Hum Reprod. 2017 Nov 1;32(11):2234-2242. doi: 10.1093/humrep/dex285. PMID 29025055
- [Background] Shapiro DB, Pappadakis JA, Ellsworth NM, Hait HI, Nagy ZP. Progesterone replacement with vaginal gel versus i.m. injection: cycle and pregnancy outcomes in IVF patients receiving vitrified blastocysts. Hum Reprod. 2014 Aug;29(8):1706-11. doi: 10.1093/humrep/deu121. Epub 2014 May 20. PMID 24847018
- [Background] Paulson RJ, Collins MG, Yankov VI. Progesterone pharmacokinetics and pharmacodynamics with 3 dosages and 2 regimens of an effervescent micronized progesterone vaginal insert. J Clin Endocrinol Metab. 2014 Nov;99(11):4241-9. doi: 10.1210/jc.2013-3937. Epub 2014 Feb 25. PMID 24606090